CLINICAL TRIAL: NCT07292090
Title: Yogabaserade övningar Som Kompletterande Behandling Vid migrän Och/Eller klusterhuvudvärk YOURHEAD - a Pilot Study
Brief Title: Yogabased Movements for Primary Headaches (Migraine and/or Cluster Headache) - YOURHEAD - a Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Marian Papp, Principal investigator, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNR 2025-06544-01 headache
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-10

CONDITIONS: Cluster Headache - Episodic and Chronic; Migraine Headache; Migraine Headache, With or Without Aura; Migraine in Adults; Migraine Headaches; Cluster Headaches and Other Trigeminal Autonomic Cephalgias; Migraine Disorder
Keywords: yogabased exercises; body-awareness exercises; breathing exercises; tele-health; webb based intervention
MeSH Terms: conditions — Cluster Headache; Bronchiolitis Obliterans Syndrome; Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Yogabased movements weekly (online live or face to face) for primary headaches
  Interventions: Other: Intervention yogabased movements

INTERVENTIONS:
Other: Intervention yogabased movements — Yogabased movements weekly (online) or face to face for primary headaches"

SUMMARY:
Migraine and/or Cluster Headache: Study Overview

**Background:** Migraine and cluster headache are two primary headache disorders that significantly impact quality of life and functionality in those affected. According to the WHO's recurring burden of disease reports, migraine is among the neurological conditions responsible for the highest number of years lost due to illness. The headaches associated with migraine and cluster headache range from moderate to severe and cause great suffering. Available treatments do not work for everyone and are often associated with adverse side effects. Physical activity has been shown in several studies to have a positive effect on headache. Given the high prevalence of mental health issues, stress, and sleep problems within this patient group, relaxation and low-intensity exercise such as yoga-based movements (YB) could potentially help individuals improve sleep and well-being, while also providing some preventive effect on headaches.

**Hypothesis:**

Individuals with severe migraine or cluster headache have a strong need for new treatment options. Alternative therapies such as yoga-based exercises, when combined with standard medical treatment as per clinical guidelines, may positively impact:

1. Headache symptoms
2. Sleep quality
3. Overall life quality

**Purpose and Goals:** This pilot study aims to evaluate the feasibiiity of a web-based yoga or live face to face (FTF) intervention in individuals suffering from severe primary headaches-mainly chronic migraine and/or cluster headache. The study will assess the effect of YB on health-related quality of life, with a focus on sleep quality and mental health as depression and anxiety. A secondary objective is to analyze changes in headache frequency, intensity, and duration associated with primary headache conditions. The pilot study will follow later on with a RCT study (will be registered later). The RCT study will have a comparison group to conventional treatment.

**Relevance for the Patient Group:** The core objective of the project is to determine whether yoga-based exercises can serve as a complementary treatment to enhance quality of life and health in patients with severe primary headache. To ensure equal healthcare access, this intervention will be delivered in digital format and/or FTF to optimize availability and expand care for individuals with primary headache disorders. These efforts aim to improve life quality and well-being in a vulnerable patient population. Headache conditions often affect individuals in their most productive years, and many live with symptoms for decades. Both work and private life are frequently disrupted, resulting in sick leave and social isolation. Close relatives are also affected, as those suffering from headaches require more recovery time to cope with daily life. With this proposed project, we aim to use physical yoga, rooted in holistic traditional medicine, to help individuals with severe primary headache achieve better physical and mental health-particularly improved sleep quality, which in turn enhances overall life quality.

DETAILED DESCRIPTION:
Current Situation

Migraine and cluster headache are two neurological conditions characterized by recurrent attacks of severe headache. Approximately 14% of the population is estimated to suffer from migraines, while cluster headaches have a prevalence of around 0.1%. The phenotype is marked by unilateral headache attacks lasting approximately 15 minutes to three hours for cluster headache and three hours to three days for migraine. Acute treatment for migraines and cluster headaches typically involves triptans or oxygen therapy to break the attacks, and prophylactic treatment when needed.

Studies have shown that individuals with headaches experience significant impacts on quality of life and often suffer from mental health issues. Research from Karolinska Institutet and the Headache Centre in Copenhagen has demonstrated sleep disturbances among individuals with cluster headaches. Sleep-related diagnoses are also frequently reported in individuals with migraine, and migraine is more prevalent among shift workers compared to non-shift workers. Collectively, these studies indicate a strong connection between sleep problems, mental health, and headache.

The disease burden in high-frequency migraine, chronic migraine, and cluster headache is substantial, and additional alternative treatments are needed alongside standard pharmaceutical therapies. Individuals with these headache types report higher sick leave rates than the general population, and cluster headache sufferers with concurrent mental health issues show increased prevalence for long-term sick leave and disability pension.

Role of Yoga-Based Exercises (YB)

Yoga-based exercises have gained attention in healthcare and are used as complementary treatments for various conditions. Reviews and meta-analyses show effects on stress symptoms, mental states such as sleep disturbances and depression. Web-based yoga interventions have also improved sleep and stress, as well as chronic neck and back pain. Improvements have been observed in endothelial function and inflammation markers.

A review article from China indicates that physical yoga (similar to the planned intervention) appears to reduce headache intensity, duration, and frequency. Previous studies show reductions in migraine headache following yoga interventions, and smaller Indian studies report effects on headache intensity and quality of life in migraine. Research in Western contexts is limited and studies conducted in India tend to show more positive results-possibly due to higher treatment dosages or contextual influences, including placebo or Hawthorne effects.

The American Migraine Foundation recommends yoga-based exercises as a complementary treatment for stress reduction and migraine symptom management, as stress is a common migraine trigger. There is currently no research on yoga-based interventions for cluster headaches, and only a few published studies on migraines.

Traditional Medical Practices

Indian traditional medicine recommends specific exercises (e.g., inversions) for treating headaches, high blood pressure, and improving sleep quality and insomnia. Inversions appear to activate deep brain regions related to sleep and have a calming effect. Sleep disorders often trigger migraines and vice versa. Melatonin rhythms, which may be unstable in headache conditions, often stabilize following yoga-based interventions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed chronic migraine and/or cluster (Hortons) headache
* Men and women 18-65 years
* Diagnosed with chronic/high frequency migraine (≥15 headache days/month with at least ≥8 with migraine)
* Diagnosed with chronic cluster head ache (i.e shorter remission than 3 months per year), diagnosed according to ICHD-III criteria.
* Ability to perform yoga based moments and to give consent.
* Internet connection with computer/ipad/mobile to perform digitally/tele-health instructions

Exclusion Criteria:

* Recent or planned operations during the last 6 weeks
* Drug dependence, alcohol dependence, mental disorders as psychosis, bipolar disorder, anxiety as PTSD etc)
* Parallel enrollment in other clinical trails
* Unmedicated high blood pressure, heart disease as heart failure
* Non Swedish speaking
* Not able to perform low intensity exercise at home or FTF (face to face) - both online or live.
* Participants unsure to participate due to drug addiction or other causes
* Disorientation and not able to inform regarding other serious conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sleep quality using insomnia severity scale (ISI) | Baseline and 8-12 weeks after the intervention, follow up after 3 and 6 months
  Total score from 0-28 - a score of 0-7 no clinical insomnia, 8-14 no insomnia, 15-21 clinical insomnia moderate, 22-28 clinical insomnia severe
Quality of life - headache intensity scale (HIT-6) | Baseline and 8-12 weeks after the intervention and follow-up after 3 and 6 months
  Total score between 36-78, low scores indicates high quality of life
Karolinska Sleep questionnarie (KSQ) - subjective sleepiness | Baseline and 8-12 after the intervention as well as follow-up 3 months and 6 months
  KSQ includes 18 questions - on a 6 graded likert scale between 0-5, where 0 = never and 5 = always. Higher scores means more sleep problems. Each domain is calculated with a mean, sleep quality 4 questions, problem waking 3 questions, sleep apnea (breath pause - andningsuppehåll) - 3 questions, sleepiness/tiredness - 6 questions. One is not using total scores for the KSQ. It is also possible to calculate index-value for insomnia and sleep apnea.
  There are cut-off values to compare with a healthy population or other studies with the same disorder. There are cut-offs for KSQ for normal swedish population but also using the 90:e percentile for a swedish population (different for men and women)
Dysfunctional Beliefs and attitudes about sleep (DBAS-10) | Baseline and after 8-12 weeks of intervention and follow-up after 3 and 6 months
  Measures sleep related cognitions in a VAS-scale. The scale identifies specific, irrationell and affective thoughts that can disturb insomnia and evaluated sleep related cognitions. Factor I (5 items) was labeled Beliefs about the Immediate Negative Consequences of Insomnia. Factor II (3 items) was labeled Beliefs about the Long-term Negative Consequences on Insomnia. Factor III was labeled Beliefs about the Need for Control Over Insomnia (2 items). Administration time 10 minutes

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Baseline and after intervention of 8-12 weeks and follow-up after 3 and 6 months
  HADS Hospital Anxiety and Depression Scale (HADS) is a self-report questionnaire designed to assess anxiety and depression levels in individuals, particularly in non-psychiatric hospital settings. Structure: The questionnaire consists of 14 items, divided into two subscales: HADS-A for anxiety and HADS-D for depression. HADS uses a 4-point Likert scale (0 = not at all, 3 = most of the time), with separate scores for anxiety and depression subscales (0-21 each). Total scores range from 0 to 42, with higher scores indicating greater symptom severity. Cut-off scores for interpretation include:
  0-7: Normal. 8-10: Mild. 11-21: Moderate to severe.
Perceived stress scale (PSS-10) | Baseline and after 8-12 week intervention, follow-up after 3 and 6 months
  The interpretation of PSS-10 scores is not diagnostic but provides a general sense of where a person falls on the spectrum of perceived stress. Generally, a score between 0-13 is considered low stress, 14-26 is moderate stress, and 27-40 is high stress.
Generalized Anxiety Disorder scale (GAD-7) | Baseline and 8-12 after the intervention as well as follow-up 3 months and 6 months
  The GAD-7 score helps assess the severity of anxiety symptoms, with scores ranging from 0 to 21 indicating varying levels of anxiety severity.
  0 - 4: No to Minimal Symptoms - Indicates little to no anxiety symptoms. 5 - 9: Mild Symptoms - Suggests mild anxiety that may not significantly impact daily functioning.
  10 - 14: Moderate Symptoms - Indicates moderate anxiety, which may affect daily activities and quality of life.
  15 - 21: Severe Symptoms - Reflects severe anxiety that likely requires clinical intervention and support.
  Clinical Relevance A score of 10 or higher may indicate a preliminary diagnosis of Generalized Anxiety Disorder (GAD).
Headache diary - frequency, intensity and duration | Baseline and after the 8-12 weeks after the intervention and follow-up after 3 and 6 months
  Headache frequency (number of days a month and number of attacks per day), headache intensity/pain using a VAS-scale, head ache duration (number of hours/minutes during an attack).
Nijmegen Dysfunctional breathing scale | Baseline and after 8-12 weeks after the intervention and 3 and 6 months follow-up
  The Nijmegen Questionnaire (often called the Nijmegen Dysfunctional Breathing Scale) is a validated screening tool designed to identify symptoms of dysfunctional breathing, particularly hyperventilation syndrome. It consists of 16 symptom items scored on a 0-4 scale, with higher scores indicating greater respiratory distress. A total score above 19-23 suggests clinically relevant breathing dysfunction. 16 items covering common symptoms such as chest pain, dizziness, blurred vision, shortness of breath, and feelings of tension.
  Each item is rated on a 5-point Likert scale: 0 = Never, 1 = Rarely, 2 = Sometimes, 3 = Often, 4 = Very often.
  * 19 points: Indicates possible dysfunctional breathing or hyperventilation.
  * 23 points: Stronger indication of hyperventilation syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Huddinge, Sweden